CLINICAL TRIAL: NCT00430014
Title: An Open-Label Study of the Safety and Efficacy of Atiprimod Treatment for Patients With Advanced Cancer
Brief Title: Study of Atiprimod Treatment for Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Withdrew
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Callisto Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0913
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Relapsed; Atiprimod; Guanylyl cyclase receptor antagonist
MeSH Terms: conditions — Recurrence | interventions — azaspirane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atiprimod (Experimental)
  Interventions: Drug: Atiprimod

INTERVENTIONS:
Drug: Atiprimod — Starting Dose of 60 mg/day orally for 14 days of 28 day cycle.

SUMMARY:
Primary Objectives:

The primary objectives of this study are to identify the maximum tolerated dose (MTD) and to evaluate the safety of atiprimod when given in doses starting at 60 mg/day and ranging to 360 mg/day, or the MTD, whichever is lower, in patients with advanced cancer.

Secondary Objectives:

The secondary objectives of this study are to measure the pharmacokinetics of atiprimod and to evaluate the efficacy of atiprimod treatment in patients with advanced cancer, and to compare the pharmacokinetics of atiprimod tablets and capsules at the starting dose, with the intent of switching to capsules for the dose escalation if the capsules pose no safety issues.

DETAILED DESCRIPTION:
Atiprimod was shown to slow or stop the growth of several human tumor cell lines in laboratory studies. Researchers believe it may have the same effect on tumor cells in patients with advanced cancer.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. At the screening visit, you will be asked questions about your medical history and any medications you use. You will be asked questions about your ability to carry out everyday activities (performance status). You will have a complete physical exam, including measurement of your vital signs (blood pressure, pulse, breathing rate, and temperature), routine blood (about 1 teaspoon) and urine tests, and an electrocardiogram (ECG--a test to measure the electrical activity of the heart).

You will have a neurological exam, which will include a series of questions and tasks (such as walking, talking, and touching your nose). The interview will take about 20 minutes to complete. Additionally, the study doctor will test your reflexes by tapping your arms, knees, and the bottom of your feet with a rubber triangle-shaped end of a special instrument that looks like a little hammer. The study doctor will also test your ability to sense light touch and pinprick, and will check your eyes with a special light source (ophthalmoscope). You will be asked questions about your physical, social/family, emotional, and functional well-being, as well as additional concerns you may have regarding numbness, tingling, discomforts, and difficulties you may be having. The interview will take about 10 minutes to complete.

The tumor will be measured by tests that are normally used to check the extent of disease in patients with the same type of cancer. This may include x-rays, MRIs, CT scans, or bone marrow biopsies. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must also have a negative pregnancy test in order to participate in this study.

If you complete all of the screening tests and are eligible to participate in the study, you will be scheduled to return to the clinic within 14 days, for baseline testing and the start of treatment (Day 1). You will be asked questions about your medical history and the medications you used since the last visit. You will have a physical exam, including measurement of your vital signs, and routine blood tests (about 1 teaspoon). A blood sample (roughly less than half of a teaspoon) will also be drawn for pharmacokinetic (PK) testing. PK testing is used to measure the amount of atiprimod in your blood. This first blood sample will be your "baseline" PK sample, and the drug level in later blood samples will be compared to it.

You will be assigned to one of 8 specific dose levels of atiprimod, based on when you entered the study; however, your dose level may be lowered if you experience increased blood levels of AST and ALT (liver function tests used to monitor for possible liver inflammation). Your assigned dose level will decide how many tablets or capsules of atiprimod you will take for each dose. The first group of 3 patients will receive atiprimod tablets at the lowest dose level for 14 days, followed by 14 days off drug. If no serious side effects occur, the next 3 patients will receive atiprimod capsules at the lowest dose level. If no serious side effects occur, the next 3 patients will receive atiprimod capsules at the next higher dose level and capsules will be used for the rest of the study (tablets will only be used for the first group of 3 patients). If 1 of the 3 patients experiences a serious side effect, the next 3 patients will be given the same dose (rather than the next higher dose) to further evaluate safety at that dose. If no serious side effects occur, the next 3 patients will receive the next higher dose. Each new dose level will be tested in this way, until the highest dose level (8th dose level) is reached or until serious side effects occur, in which case the dose will not be raised any higher.

During the study, you will take your dose of atiprimod orally (by mouth) in tablet or capsule form once a day for 14 days, followed by 14 days with no atiprimod treatment. These 28 days (4 weeks) will make up one treatment "cycle." If you do not experience a serious side effect that forces your doctor to remove you from study, and your cancer is stable or shrinking after 2 months of treatment, you will be eligible to continue on atiprimod treatment for up to 1 year (a total of 12 cycles). If you experience increased blood levels of AST and ALT, and these levels return to normal within 7 days of completing the treatment cycles, you may be eligible to continue atiprimod treatment, but at a lower dose level and on a modified schedule (atiprimod once a day for 7 days, followed by 7 days off atiprimod). You should take the atiprimod in the morning at about the same time each day. You should not eat food for at least 2 hours before and 2 hours after taking atiprimod. You should drink 1 - 2 glasses of water (preferred) or orange juice, soda, tea, or coffee during the 2 hours before and 2 hours after taking your daily dose of atiprimod, and you may drink water (preferred) or orange juice, soda, tea, or coffee during the 2-hour period after taking your daily dose of atiprimod.

After your baseline testing, you will be given your first dose of atiprimod. During the first 8 hours after your first dose of atiprimod, you will be watched for any side effects that might occur. You will have several blood samples taken during this period for PK testing. About a quarter of a teaspoon of blood will be drawn 30 minutes after your first dose, then again at 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, and 8 hours after your first dose, for a total of 2 teaspoons of blood drawn. After these blood collections, you will go home. You will be given a study diary for recording any other medications you take and how much you take, as well as any side effects that you experience. You will also be asked to record the type and amount of beverage consumed during the 2-hour period before taking atiprimod and the 2-hour period after taking atiprimod. You will be required to keep this diary up to date during your entire participation on study, and you must bring it to every study visit.

You will return to the clinic 24, 48, and 72 hours after your first dose (Study Days 2, 3, and 4). You will be asked questions about your medical history and the medications you used since the last visit. You will have a physical exam, including measurement of your vital signs, routine blood (about 1 teaspoon), and an ECG. The ECG will only be done on Day 2 (not on Days 3 and 4). A blood sample (less than half of a teaspoon) will be drawn for PK testing. You will be given your daily dose of atiprimod.

Before you leave the clinic on Study Day 4, you will be given enough atiprimod to last until the next visit (in other words, through Study Day 6). You will be instructed to not eat food for at least 2 hours before or 2 hours after taking atiprimod, and to take the atiprimod in the morning at the same time each day. You will also be instructed to drink 1 - 2 glasses of water (preferred) or orange juice, soda, tea, or coffee during the 2 hours before and 2 hours after taking your daily dose of atiprimod. You will be given a diary for recording when you take the atiprimod, the type and amount of beverage consumed during the 2-hour period before taking atiprimod and the 2-hour period after taking atiprimod, other medications that you take, and any side effects that you experience.

You will be asked to return to the clinic for tests once a week during the first cycle of treatment (Days 7, 14, 21, and 28). You will take the atiprimod doses on Days 5-14 at home as instructed, except for the 2 days during this period that you are scheduled to return to the clinic (Study Days 7 and 14). These 2 doses will be given to you at the clinic. Before you leave the clinic on Study Day 7, you will be given enough atiprimod to last until the next visit (Study Day 14).

During these first four weekly visits (Study Days 7, 14, 21, and 28), you will have several tests performed. During each visit, you will be asked questions about your medical history and the medications you used since the last visit. You will be asked questions about the doses of atiprimod you have taken on your own (number of tablets or capsules taken at each dose, time each dose was taken, if you ate food or drank something other than water, orange juice, soda, tea, or coffee during the 2 hours before or after taking study drug, and the number of glasses of water, orange juice, soda, tea, or coffee that you drank during this 4-hour period). You will have a physical exam, including measurement of your vital signs, routine blood (about 1 teaspoon) and urine tests. You will have an ECG at Day 28 only (not on Days 7, 14, or 21). You will also have a neurological exam. You will be asked questions about your physical, social/family, emotional, and functional well-being, as well as additional concerns you may have regarding numbness, tingling, discomforts, and difficulties you may be having.

You will have several PK blood samples taken at your Day 14 visit. About a quarter of a teaspoon will be taken 30 minutes after you take the atiprimod dose at your Day 14 visit, and then again at 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, and 8 hours after that same dose, for a total of 2 teaspoons of blood drawn. You will also be instructed to return to the clinic 24, 48, and 72 hours after your Day 14 visit for a single blood collection. Less than a quarter of a teaspoon of blood will be collected at each of these 3 visits. A single blood collection (about half of a teaspoon) will also be taken at your Day 7, Day 21 and Day 28 visits for PK testing.

At your Day 28 visit, you will also have the size of the tumor measured using x-rays, MRIs, or CT scans, as before. Women who are able to have children will have a blood pregnancy test.

After the first cycle, you will return to the clinic for evaluation once a month at the end of each cycle that you are eligible for treatment. If you do not experience a serious side effect that forces your doctor to remove you from study, and your cancer is stable or shrinking after 2 months of treatment, you will be eligible to continue on atiprimod treatment for up to 1 year (a total of 12 cycles).

At each monthly study visit, you will be given enough atiprimod to last until your next clinic visit (Week 4 of next cycle). You will be given a diary for recording when you take the atiprimod, the type and amount of beverage consumed during the 2-hour period before taking atiprimod and the 2-hour period after taking atiprimod, other medications that you take, and any side effects that you experience. During these monthly visits, you will have several tests performed. You will be asked questions about the doses of atiprimod you have taken on your own. You will have a physical exam, including measurement of your vital signs, routine blood (about 1 teaspoon) and urine tests, and an ECG. You will have a neurological exam. You will be asked questions about your physical, social/family, emotional, and functional well-being, as well as additional concerns you may have regarding numbness, tingling, discomforts, and difficulties you may be having. A single blood collection (less than half of a teaspoon) will be taken for PK testing. Your tumor will be measured using the same kinds of scans as before. Women who are able to have children will have a blood pregnancy test.

If you experience increased blood levels of AST and ALT, and these levels return to normal within 7 days of completing the treatment cycle, you may be eligible to continue atiprimod treatment, but at a lower dose level and on a modified schedule. If you do receive a modified schedule of atiprimod, you will return to the clinic for an additional evaluation on Week 2 (Day 14) of the modified cycle (in addition to the evaluation that you will have at the end of the cycle). This evaluation will include the same tests done at the monthly visits, except that your tumor will not be measured and you will not have a pregnancy test.

Extra visits, tests, and/or procedures may be done at any time during this research study, if the doctor thinks they are in your best interest.

You will be taken off study if the disease progresses, intolerable side effects occur, or you do not follow study guidelines for participation.

One month after your last treatment cycle, you will return to the clinic for a follow-up evaluation. You will be asked questions about your ability to carry out everyday activities (performance status). You will be asked questions about your medical history and the medications you used since the last visit. You will have a physical exam, including measurement of your vital signs, routine blood (about 1 teaspoon) and urine tests, and an ECG. You will have a neurological exam. You will be asked questions about your physical, social/family, emotional, and functional well-being, as well as additional concerns you may have regarding numbness, tingling, discomforts, and difficulties you may be having. A single blood collection (less than half of a teaspoon) will be taken for PK testing. Women who are able to have children will have a blood pregnancy test.

This is an investigational study. Atiprimod is authorized by the FDA for research only. About 61 individuals will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histological proof of advanced cancer and must have failed or relapsed following standard therapy or have no standard therapy available.
2. Patient must have an estimated life expectancy of at least 12 weeks.
3. Patient must have measurable or evaluable disease.
4. Patient has an ECOG (Zubrod) performance status of 0 to 2.
5. Age >/= 13 years at the time of signing informed consent.
6. All necessary screening evaluations for determining eligibility must be obtained within 14 days prior to the first dose of study drug except for measurement of disease extent, which can be obtained within 28 days prior to the first dose of study drug.
7. Patient must be able to adhere to the study visit schedule and other protocol requirements.
8. Patient must understand and voluntarily sign an informed consent document.
9. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

Exclusion Criteria:

1. Renal insufficiency (serum creatinine levels >/= 2 times the upper limit of normal).
2. Concomitant radiotherapy, chemotherapy, or other investigational agents/therapies.
3. Peripheral neuropathy of Grade 3 or greater assessed by a directed neurologic examination, including light touch, pinprick, proprioception, and deep tendon reflexes of the upper and lower extremities; and questioning for symptoms of paresthesia and numbness (FACT/GOG-Ntx: Appendix D).
4. Patients with evidence of clinically significant mucosal or internal bleeding. (For example, a decrease in hemoglobin of greater than 1.5 gm will be considered clinically significant.)
5. Patients with a platelet count < 50,000 cells/mm^3.
6. Patients with an absolute neutrophil count (ANC) of < 1000 cells/mm^3.
7. ALT/SGPT or AST/SGOT levels >/= 2 times the upper limit of normal (ULN) except in patients with documented hepatic metastases.
8. Total bilirubin > 2 times the ULN.
9. Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study. Such examples include infection requiring hospitalization and psychiatric health which would make compliance understanding difficult.
10. Clinically relevant active infection or serious co-morbid medical conditions such as recent (</6 months) MI, unstable angina, difficult to control CHF, uncontrolled HTN, difficult to control cardiac arrhythmias, COPD or chronic restrictive pulmonary disease, and cirrhosis. Examples of uncontrolled HTN and difficult to control cardiac arrhythmias include situations in which patients still have the problem while on medication or patients who have required > two medication changes in the last 6 months in order to control the problem, or cardiac patients with a NYHA classification of > Class II.
11. If WCBP, pregnant, lactating, or not using adequate contraception.
12. As atiprimod is a potent inhibitor of CYP2D6 (a chemical that is produced naturally by the body that processes and eliminates certain types of chemicals), patients taking drugs that are substrates of CYP2D6 (e.g., beta blockers, antidepressants, and antipsychotics; see Appendix G) will be excluded from the study.
13. Received any form of radiotherapy, chemotherapy, or other investigational agents/therapies within 30 days prior to the first dose of study drug.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Atiprimod | With each 28 day (4 week) cycle

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org